CLINICAL TRIAL: NCT05306028
Title: Administration of Metformin and Insulin to Pancreatic Cancer Related Diabetes Mellitus (Type 3c)
Brief Title: Metformin and Insulin to Pancreatic Cancer Related Diabetes (Type 3c)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCA199-2
Record Dates: First submitted 2022-03-03; First posted 2022-03-31 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Pancretic Cancer; Diabete Mellitus
Keywords: blood glucose; metformin; insulin
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metformin or insulin treatment (Experimental)
  Interventions: Drug: Metformin or insulin treatment

INTERVENTIONS:
Drug: Metformin or insulin treatment — 1. For patients with new-onset diabetes Fasting blood glucose 7-10 mmol/L, metformin 2 g/day, BID, PO; Fasting blood glucose 10-14 mmol/L, metformin 1 g/day, BID, PO, Novolin 30R Penfil 12 U before breakfast, 8 U; Fasting blood glucose > 14 mmol/L, metformin 1 g/day, BID, PO, Novolin 30R Penfil 16 U before breakfast, 10 U; Adjusting insulin dosage according to the monitor of fasting blood glucose.
  2. For patients with history of diabetes Adjusting metformin or insulin dosage according to the monitor of fasting blood glucose.

SUMMARY:
About 80% of patients with pancreatic adenocarcinoma have aberrant fasting blood glucose at the time of diagnosis. The consistent association between pancreatic cancer and diabetes mellitus has long been recognized and even been termed as "chicken and egg". Many reports have found that pancreatic cancer can result in diabetes, which is called type 3c diabetes. New-onset diabetes is commonly observed in pancreatic cancer patients and has been considered as a potential screening sign. Moreover, diabetes has been found as a predictor of poor outcome in pancreatic cancer.

Pancreatic cancer cells have a strong dependence on glucose and they are well-known for their sweet teeth. High glucose is associated with impaired immunologic reaction, intolerability to chemotherapy, radiotherapy and other major treatments, an increased risk of pancreatic surgery. Given the linkage between pancreatic cancer and diabetes or high blood glucose, a clinical trial is needed to validate the effect of metformin and insulin on regulating blood glucose in type 3c diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed content obtained prior to treatment
* Age ≥ 18 years and ≤ 80 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must have histologically confirmed pancreatic adenocarcinoma
* History of diabetes mellitus, or newly diagnosed diabetes mellitus according to the American Diabetes Association criteria
* The expected survival after surgery ≥ 3 months

Exclusion Criteria:

* Active second primary malignancy or history of second primary malignancy
* Patients who have received any form of anti-tumor therapy including surgery, chemotherapy, radiotherapy, interventional chemoembolization, radiofrequency ablation, and molecular targeted therapy
* Inflammation of the digestive tract, including pancreatitis, cholecystitis, cholangitis, etc
* Pregnant or nursing women
* Patients who are unwilling or unable to comply with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood glucose control rate | 1 week
  Blood glucose control rate before and after anti-diabetic administration

SECONDARY OUTCOMES:
HbA1C control rate | 1 week
  HbA1C control rate before and after anti-diabetic administration

OTHER OUTCOMES:
Change in serum Carbohydrate Antigen 19-9 (CA19-9) From Baseline to Day 8. | 1 week
  Change of tumor biomarkers before and after anti-diabetic administration.Patients will collect CA19-9 values on the day of enrollment and on day 8.
Overall survival，OS | At the end of Cycle 1 (each cycle is 28 days)
  OS of subjects from recruiting to the time of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sharma A, Kandlakunta H, Nagpal SJS, Feng Z, Hoos W, Petersen GM, Chari ST. Model to Determine Risk of Pancreatic Cancer in Patients With New-Onset Diabetes. Gastroenterology. 2018 Sep;155(3):730-739.e3. doi: 10.1053/j.gastro.2018.05.023. Epub 2018 Jun 11. PMID 29775599
- [Background] Pannala R, Basu A, Petersen GM, Chari ST. New-onset diabetes: a potential clue to the early diagnosis of pancreatic cancer. Lancet Oncol. 2009 Jan;10(1):88-95. doi: 10.1016/S1470-2045(08)70337-1. PMID 19111249
- [Background] Bragg F, Holmes MV, Iona A, Guo Y, Du H, Chen Y, Bian Z, Yang L, Herrington W, Bennett D, Turnbull I, Liu Y, Feng S, Chen J, Clarke R, Collins R, Peto R, Li L, Chen Z; China Kadoorie Biobank Collaborative Group. Association Between Diabetes and Cause-Specific Mortality in Rural and Urban Areas of China. JAMA. 2017 Jan 17;317(3):280-289. doi: 10.1001/jama.2016.19720. PMID 28114552
- [Background] Yuan C, Rubinson DA, Qian ZR, Wu C, Kraft P, Bao Y, Ogino S, Ng K, Clancy TE, Swanson RS, Gorman MJ, Brais LK, Li T, Stampfer MJ, Hu FB, Giovannucci EL, Kulke MH, Fuchs CS, Wolpin BM. Survival among patients with pancreatic cancer and long-standing or recent-onset diabetes mellitus. J Clin Oncol. 2015 Jan 1;33(1):29-35. doi: 10.1200/JCO.2014.57.5688. Epub 2014 Nov 17. PMID 25403204